CLINICAL TRIAL: NCT02511301
Title: Circadian Thermal Sensing for the Detection of Breast Disease as a Supplemental Cancer Screening System
Brief Title: Circadian Thermal Sensing to Detect Breast Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyrcadia Health (Industry)
Collaborators: Stanford University (Other); Salesforce (Unknown); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CH001
Record Dates: First submitted 2015-06-18; First posted 2015-07-30 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Early-Stage Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyrcadia CBR™ Device (Experimental): Cyrcadia CBR™ device, including adhesive patches on both breasts connected to a small recorder, is placed on the study subject for 2 to 24 hours. After the test period, the CBR™ will be removed and the data will be downloaded to a central site for analysis.There are no interventions after the CBR™ is removed from the Study Subject
  Interventions: Device: Cyrcadia CBR™ device placement for abnormality screening

INTERVENTIONS:
Device: Cyrcadia CBR™ device placement for abnormality screening — Cyrcadia CBR™ device, including adhesive patches on both breasts connected to a small recorder, is placed on the study subject for 2 to 24 hours. After the test period, the CBR™ will be removed and the data will be downloaded to a central site for analysis. There are no interventions after the CBR™ is removed from the Study Subject.

SUMMARY:
The purpose of this study is to determine if Cyrcadia's Circadian Biometric Recorder (CBR™), which is attached to soft biometric patches worn on the body, can improve early breast cancer detection along with mammography or as a stand alone device.

DETAILED DESCRIPTION:
The Cyrcadia CBR™ (Circadian Biometric Recorder) includes wearable biometric patches and a detachable data recording device. The CBR™ records chronobiologic data while the patient is totally ambulatory and going about her normal daily routine. Following removal of the detachable data recording device from the wearable biometric patches, the data is transferred to a computer for analysis. The Cyrcadia CBR™ will be placed on the patient for the duration of 2 to 24 hours. There is no restriction of daily activity. The study subject is requested to sponge bathe rather than shower while wearing the device, keeping the device dry during the testing procedure. After this period, the CBR™ will be removed and the data will be transferred to a computer for analysis.

The primary endpoint of this 173 patient study is to determine the accuracy of Cyrcadia CBR™ as a supplemental screening device to mammography and ultrasound in predicting a diagnosis of breast cancer. Specific emphasis will be on the utilization of the CBR as a secondary screening device to reduce the number of biopsies currently performed on non-cancerous tissue. A secondary emphasis will be on the CBR to act as an improved screening solution over mammography specifically in those patients with dense breast parenchymal tissue.

Other endpoints of the study are:

* to determine the accuracy of Cyrcadia CBR™, including the positive predictive value, negative predictive value, false negative rate and false positive rate.
* to determine the optimal wear time for the Cyrcadia CBR™.
* to demonstrate substantial equivalent or improved results when applied to Cyrcadia original patient case study with identical advanced neural network analysis computational results.

Study subjects will be followed at 6, 12, 18, and 24 months to update their clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Women with a BI-RADS category 4 or 5 designation on mammogram
* Women with a BI-RADS category 4 or 5 designation on breast ultrasound
* Women with a BI-RADS category 4 or 5 designation on breast MRI
* Women who are willing to undergo a complete evaluation and/or biopsy procedure if recommended by the treating physician

Exclusion Criteria:

* Less than 21 years of age
* Unable to sign the consent form
* Pregnant or lactating
* Physically unable to wear the Cyrcadia CBR™ for 6 hours
* Previous mastectomy
* Any breast surgery or biopsy within the last 90 days
* Any trauma to the breast within the last 90 days
* Any biopsy or treatment for the BI-RADS category 4 or 5 abnormality
* Refusal to undergo recommended diagnostic evaluation of the BI-RADS category 4 or 5 abnormality

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Predictive Analytic Analysis (PAA) Sensitivity and Specificity | 7 to 30 days after CBR placement
  The data is analyzed using a predefined set of algorithms, referred to as Predictive Analytic Analysis (PAA) Outcome is measured by: NUMBER OF PATIENTS WHOSE INVESTIGATIVE CBR DEVISE RESULTS MATCH OF THOSE OF THE BIOPSY RESULTS.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Ellenhorn, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - El Camino Hospital, Mountain View, California
  - The Ohio State University, Stephanie Spielman Comprehensive Cancer Center, Columbus, Ohio